CLINICAL TRIAL: NCT01486875
Title: NovoMix® Start - A Multicentre, Open Label, Non-randomised, Non-interventional, Observational Safety Study in Subjects With Type 2 Diabetes Mellitus Starting NovoMix 30® Treatment
Brief Title: Observational Study of Safety of NovoMix® 30 Treatment for Type 2 Diabetes
Acronym: Start
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1721
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BIAsp 30
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted, and administered subcutaneously (under the skin) once or twice daily

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the incidence of serious adverse drug reactions when initiating insulin therapy with NovoMix® 30 in subjects with type 2 diabetes mellitus under normal clinical practice conditions in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After the physician has decided to initiate biphasic insulin aspart 30 therapy, any insulin-naïve patient with type 2 diabetes mellitus in need of improved metabolic control, as judged by the treating physician, will be able to participate
Sampling Method: Non-Probability Sample
Enrollment: 1155 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) | Week 26
Incidence of major hypoglycaemic events | Week 26

SECONDARY OUTCOMES:
Number of all hypoglycaemic events | In the 4 weeks prior to week 12 and week 26, respectively
HbA1c (glycosylated haemoglobin A1c) | Week 26
Fasting Plasma Glucose (FPG) | Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Lund, Sweden

REFERENCES:
- [Result] Berntorp K, Haglund M, Larsen S, Petruckevitch A, Landin-Olsson M; Swedish BIAsp Study Group. Initiation of biphasic insulin aspart 30/70 in subjects with type 2 diabetes mellitus in a largely primary care-based setting in Sweden. Prim Care Diabetes. 2011 Jul;5(2):89-94. doi: 10.1016/j.pcd.2011.02.003. Epub 2011 Mar 26. PMID 21440523
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com